CLINICAL TRIAL: NCT06762548
Title: Clinical Study of DA-007 for the Treatment of Chemotherapy Induced Alopecia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Applied Biology, Inc. (Industry)
Collaborators: Daniel Alain, Inc. (Unknown); Follea International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DA-007-CIA
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Chemotherapy Induced Alopecia; Chemotherapy Side Effects
Keywords: Chemotherapy Induced Alopecia; Chemotherapy Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DA-007 (Active Comparator): Topical DA-007 Solution
  Interventions: Drug: DA-007
- Placebo (Placebo Comparator): Topical Placebo Solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DA-007 — Topical α1 agonist combination of Phenylephrine + Tyramine + Synephrine
  Arms: DA-007
Drug: Placebo — Topical placebo solution
  Arms: Placebo

SUMMARY:
Clinical Study of DA-007 As a Treatment for Chemotherapy Induced Alopecia

DETAILED DESCRIPTION:
Chemotherapy induced alopecia (CIA) is a common adverse event of oncological treatment. The significant psychological burden of CIA, particularly in women, leads some (~8%) to reject life saving therapeutic regimens. Several studies have demonstrated the effectiveness of scalp vasoconstriction as a prophylactic treatment for CIA. Recently, US Food and Drug Administration (FDA) approved a scalp-cooling device as a prophylactic treatment for CIA. Scalp cooling results in reduced local blood perfusion and consequently reduced chemotherapeutic agents reaching the hair follicle niche; however, scalp cooling requires prolongation of the time required to attend the chemotherapy unit (>2 hrs) as well as common adverse events including intolerance to cold. A previous study demonstrated that the α1 agonist, phenylephrine hydrochloride, applied topically can penetrate the scalp and bind α1 receptors. As such, a topically applied α1 agonist would reduce scalp blood perfusion. A novel formula (DA-007), containing an α1 agonist, that can also penetrate the scalp and bind α1 receptors. The aim of the study is to test the hypothesis that DA-007 can reduce scalp blood perfusion and thus reduce hair loss due to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stage I or stage II breast cancer
* Scheduled but not begun, at least 4 cycles of taxane and/or anthracycline-based chemotherapy.
* Ages 18-65
* Able to give informed consent

Exclusion Criteria:

* Resting blood pressure outside the range of 105-140/ 55-99
* Uncontrolled or severe hypertension
* Female pattern hair loss or hair loss disorder
* Folliculitis
* Scalp psoriasis
* Seborrheic dermatitis
* Inflammatory scalp conditions such as lichen planopillaris
* Subjects wearing wigs prior to chemotherapy
* Use of MAO inhibitors
* Unable to provide consent or make allotted clinical visits

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 140 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2026-09-11 (Estimated); Study Completion 2026-11-06 (Estimated)

PRIMARY OUTCOMES:
Prevention of Hair Loss (Common Terminology Criteria for Adverse Events V5.0) | Week [0,12]
  Amount of hair loss during chemotherapy treatment measured by the Common Terminology Criteria for Adverse Events (CTCAE) V5.0. The Common Terminology Criteria for Adverse Events is a common terminology developed by the National Cancer Institute to describe and grade adverse events related to cancer therapy.

SECONDARY OUTCOMES:
Hair Re-Growth Post Treatment (Common Terminology Criteria for Adverse Events V5.0) | Week [12, 24]
  Amount of hair re-growth post chemotherapy treatment measured by the Common Terminology Criteria for Adverse Events (CTCAE) V5.0. The Common Terminology Criteria for Adverse Events is a common terminology developed by the National Cancer Institute to describe and grade adverse events related to cancer therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Andy Goren, MD, Study Director — University of Rome G. Marconi
Locations (1):
- University of Rome ("G. Marconi"), Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fahl WE. Complete prevention of radiation-induced dermatitis using topical adrenergic vasoconstrictors. Arch Dermatol Res. 2016 Dec;308(10):751-757. doi: 10.1007/s00403-016-1691-2. Epub 2016 Oct 4. PMID 27704205
- [Background] Soref CM, Fahl WE. A new strategy to prevent chemotherapy and radiotherapy-induced alopecia using topically applied vasoconstrictor. Int J Cancer. 2015 Jan 1;136(1):195-203. doi: 10.1002/ijc.28961. Epub 2014 May 16. PMID 24811525